CLINICAL TRIAL: NCT02743780
Title: A Three Part, First-in-human, Randomized, Double-masked, Placebo-Controlled, Safety, Tolerability and Early Efficacy Study of MGV354 in Healthy Subjects and in Patients With Ocular Hypertension or Glaucoma
Brief Title: A Three Part Study of MGV354 in Ocular Hypertension or Glaucoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Collaborators: Novartis Institute for BioMedical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MGV354-2201
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-08

CONDITIONS: Ocular Hypertension; Open-Angle Glaucoma
Keywords: Ocular Hypertension; Open-Angle Glaucoma; POAG; Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MGV354 (Experimental): Part 3: MGV354 ophthalmic suspension, 1 drop in both eyes once per day for 7 days
  Interventions: Drug: MGV354 ophthalmic suspension
- Placebo (Placebo Comparator): Part 3: MGV354 placebo, 1 drop in both eyes once per day for 7 days
  Interventions: Drug: MGV354 placebo

INTERVENTIONS:
Drug: MGV354 ophthalmic suspension
  Arms: MGV354
Drug: MGV354 placebo — Inactive ingredients used as placebo comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the clinical profile of topical-ocular MGV354 merits further development for the indication of lowering intraocular pressure (IOP).

DETAILED DESCRIPTION:
Part 1 will evaluate the safety and tolerability of single ascending doses of MGV354 compared to placebo in healthy male and female subjects. Part 2 will evaluate the safety and tolerability of MGV354 in a multiple ascending dose design (two highest tolerated doses from Part 1) compared to placebo when administered for 7 days to patients with ocular hypertension or glaucoma. Part 3 will explore the safety, tolerability and efficacy of a single dose level of MGV354 (maximum tolerated dose) compared to placebo when administered for 7 days in patients with ocular hypertension or glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent.
* Part 1: 18 to 70 years of age;
* Parts 2 and 3: 18 years of age or older;
* Able to communicate well with the investigator and understand and comply with the requirements of the study;
* Body Mass Index (BMI) between 18 and 39;
* In case of contact lens wear, willing to remove lenses 30 minutes before the first assessment until the end of the study. Corrective spectacles may be worn as needed.
* Sitting vital signs (systolic and diastolic blood pressure and pulse rate) within normal ranges as specified in the protocol;
* Part 1 (Healthy Volunteers): In good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Parts 2 and 3 (Patients): Diagnosed with open-angle glaucoma or confirmed ocular hypertension; mean IOP measurements in at least one eye after washout as specified in the protocol
* Other protocol-specified inclusion criteria may apply.

Exclusion criteria:

* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes;
* History of or current presence of clinically significant ECG abnormalities or arrhythmias;
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical or breast cancer), treated or untreated, within the past 5 years;
* Known clinical history of heart failure, myocardial infarction, or stroke;
* Exposure during the four weeks preceding the Screening visit to any topical, inhaled, or systemic corticosteroids;
* Angle grade less than Grade 2 in either eye;
* Any abnormality, including corneal thickness > 620 microns, preventing reliable applanation tonometry;
* Pregnant or lactating women and women of child-bearing potential;
* Sexually active males must agree to use a condom during intercourse while taking drug and for 6 days after stopping MGV354 medication and should not father a child in this period;
* Positive HIV, Hepatitis B Ag or Hepatitis C Ab test result at Screening;
* Abnormal liver function tests;
* History or presence of impaired renal function;
* Part 1 (Healthy Volunteers): Use of any NEW prescription drugs or herbal supplements within four (4) weeks prior to initial dosing, and/or NEW over-the-counter (OTC) medication, dietary supplements (vitamins included) within two (2) weeks prior to initial dosing.
* Parts 2 and 3 (Patients): Patients with related disease condition(s) including any form of glaucoma other than open-angle glaucoma and pseudoexfoliation and/or pigment dispersion components; patients who cannot safely discontinue use of all topical ocular and/or systemic IOP-lowering medication according to protocol-specified Washout Schedule; patients with ocular diseases or conditions as specified in the protocol; patients taking certain medications as specified in the protocol;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2016-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Science Expert, NIBR, Study Director — Novartis Institute for BioMedical Research

REFERENCES:
- [Derived] Stacy R, Huttner K, Watts J, Peace J, Wirta D, Walters T, Sall K, Seaman J, Ni X, Prasanna G, Mogi M, Adams C, Yan JH, Wald M, He Y, Newton R, Kolega R, Grosskreutz C. A Randomized, Controlled Phase I/II Study to Evaluate the Safety and Efficacy of MGV354 for Ocular Hypertension or Glaucoma. Am J Ophthalmol. 2018 Aug;192:113-123. doi: 10.1016/j.ajo.2018.05.015. Epub 2018 May 24. PMID 29802818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 study centers located in the US.
Pre-assignment Details: This study was conducted in 3 parts. A separate cohort of subjects was enrolled for each part. Of the 191 subjects enrolled (Part 1, 2, and 3 combined), 79 were exited as screen failures and 14 were discontinued prior to randomization. This reporting group includes all randomized subjects. A zero indicates no intended subjects.
Groups:
- MGV354 0.01%: MGV354 ophthalmic suspension 0.01%, 1 drop in the study eye (Part 1)
- MGV354 0.03%: MGV354 ophthalmic suspension 0.03%, 1 drop in the study eye (Part 1) or 1 drop in each eye for 7 days (Part 2)
- MGV354 0.1%: MGV354 ophthalmic suspension 0.1%, 1 drop in the study eye (Part 1) or 1 drop in each eye for 7 days (Part 2 and Part 3)
- MGV354 0.3%: MGV354 ophthalmic suspension 0.3%, 1 drop in the study eye (Part 1)
- Placebo: Placebo, 1 drop in the study eye (Part 1); 1 drop in each eye for 7 days (Part 2 and Part 3)
Period: Part 1 (3 Days)
Arm/Group | MGV354 0.01% | MGV354 0.03% | MGV354 0.1% | MGV354 0.3% | Placebo
Started | 6 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2 (8 Days)
Arm/Group | MGV354 0.01% | MGV354 0.03% | MGV354 0.1% | MGV354 0.3% | Placebo
Started | 0 | 6 | 6 | 0 | 4
Completed | 0 | 6 | 6 | 0 | 4
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 3 (7 Days)
Arm/Group | MGV354 0.01% | MGV354 0.03% | MGV354 0.1% | MGV354 0.3% | Placebo
Started | 0 | 0 | 25 | 0 | 25
Completed | 0 | 0 | 24 | 0 | 25
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects who received at least one on-treatment measurement of IOP (Full Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | MGV354 0.01% | MGV354 0.03% | MGV354 0.1% | MGV354 0.3% | Placebo | Total
Number analyzed (Participants) | 6 | 12 | 36 | 6 | 37 | 97
Age, Customized [Mean (Standard Deviation); unit: years] — Population: This study was conducted in 3 parts.
  years
    Part 1: number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
    Part 1 | 31.2 (13.61) | 51.7 (15.77) | 48.5 (17.55) | 62.7 (7.74) | 50.1 (7.51) | 48.9 (15.54)
    Part 2: number analyzed (Participants) | 0 | 6 | 6 | 0 | 4 | 16
    Part 2 |  | 59.2 (7.52) | 63.3 (7.79) |  | 63.3 (6.70) | 61.8 (7.23)
    Part 3: number analyzed (Participants) | 0 | 0 | 24 | 0 | 25 | 49
    Part 3 |  |  | 65.5 (8.17) |  | 64.8 (9.92) | 65.2 (9.02)
Sex/Gender, Customized [Number; unit: participants] — Population: This study was conducted in 3 parts.
  participants
    Female, Part 1 | 0 | 5 | 4 | 6 | 5 | 20
    Male, Part 1 | 6 | 1 | 2 | 0 | 3 | 12
    Female, Part 2: number analyzed (Participants) | 0 | 12 | 36 | 0 | 37 | 85
    Female, Part 2 |  | 4 | 3 |  | 2 | 9
    Male, Part 2: number analyzed (Participants) | 0 | 12 | 36 | 0 | 37 | 85
    Male, Part 2 |  | 2 | 3 |  | 2 | 7
    Female, Part 3: number analyzed (Participants) | 0 | 0 | 36 | 0 | 37 | 73
    Female, Part 3 |  |  | 17 |  | 17 | 34
    Male, Part 3: number analyzed (Participants) | 0 | 0 | 36 | 0 | 37 | 73
    Male, Part 3 |  |  | 7 |  | 8 | 15
Intraocular Pressure (IOP) [Mean (Standard Deviation); unit: mmHg] — IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters mercury (mmHg). Only one eye (study eye) contributed to the analysis. Population: IOP analysis was pre-specified for Part 3 subjects only.
  mmHg
    Diurnal IOP: number analyzed (Participants) | 0 | 0 | 24 | 0 | 25 | 49
    Diurnal IOP |  |  | 24.69 (2.475) |  | 24.63 (2.119) | 24.66 (2.276)
    8 AM IOP: number analyzed (Participants) | 0 | 0 | 24 | 0 | 25 | 49
    8 AM IOP |  |  | 26.60 (2.289) |  | 27.33 (3.300) | 26.97 (2.844)
    10 AM IOP: number analyzed (Participants) | 0 | 0 | 24 | 0 | 25 | 49
    10 AM IOP |  |  | 24.68 (2.571) |  | 24.77 (1.976) | 24.72 (2.263)
    Noon IOP: number analyzed (Participants) | 0 | 0 | 24 | 0 | 25 | 49
    Noon IOP |  |  | 24.46 (2.842) |  | 24.21 (2.046) | 24.33 (2.445)
    4 PM IOP: number analyzed (Participants) | 0 | 0 | 24 | 0 | 25 | 49
    4 PM IOP |  |  | 24.39 (2.521) |  | 24.21 (1.939) | 24.30 (2.221)
    8 PM IOP: number analyzed (Participants) | 0 | 0 | 24 | 0 | 25 | 49
    8 PM IOP |  |  | 23.34 (2.998) |  | 22.64 (2.344) | 22.98 (2.680)

OUTCOME MEASURES:

1. Primary Outcome: Part 3: Change in Diurnal IOP (Averaged Over 8 AM, 10 AM, Noon, 4 PM, and 8 PM) From Baseline to Day 8
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in mmHg. Diurnal IOP was defined as the average of the five time points measured (8 AM, 10 AM, noon, 4 PM, and 8 PM). Baseline diurnal IOP was the average of IOP measurements obtained at the 2 eligibility visits. Change from baseline was calculated by taking the change at each time point from baseline to Day 8 and averaging the available changes. A more negative change from baseline indicates a greater improvement, i.e., a reduction of IOP. Only one eye (study eye) contributed to the analysis.
Time Frame: Baseline, Day 8
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mmHg
Groups:
- MGV354 0.1%: Part 3: MGV354 ophthalmic suspension, 1 drop in each eye for 7 days
- Placebo: Part 3: MGV354 placebo, 1 drop in each eye for 7 days
Arm/Group | MGV354 0.1% | Placebo
Number analyzed (Participants) | 24 | 25
mmHg | -0.6 (0.43) | -1.1 (0.42)

2. Primary Outcome: Part 3: Change in IOP From Baseline to Day 8 at 8 AM, 10 AM, Noon, 4 PM, and 8 PM
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in mmHg. Baseline IOP was the average of IOP measurements obtained at the 2 eligibility visits. Change from baseline was calculated by taking the change at each time point from baseline to Day 8. A more negative change from baseline indicates a greater improvement, i.e., a reduction of IOP. Only one eye (study eye) contributed to the analysis.
Time Frame: Baseline, Day 8
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | MGV354 0.1% | Placebo
Number analyzed (Participants) | 24 | 25
mmHg
  Change from Baseline (BL) at 8 AM | 0.1 (0.57) | -1.5 (0.56)
  Change from BL at 10 AM | -0.4 (0.57) | -1.5 (0.56)
  Change from BL at noon | -0.2 (0.57) | -0.2 (0.56)
  Change from BL at 4 PM | -1.2 (0.57) | -1.4 (0.56)
  Change from BL at 8 PM | -1.1 (0.57) | -0.7 (0.56)

3. Secondary Outcome: Part 3: Change From Baseline in IOP at 36 Hours and 48 Hours Post Day 7 Administration
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in mmHg. Baseline IOP was the average of IOP measurements obtained at the 2 eligibility visits. Change from baseline was calculated by taking the change at each time point from baseline to Day 8 and averaging the available changes. A more negative change from baseline indicates a greater improvement, i.e., a reduction of IOP. Only one eye (study eye) contributed to the analysis.
Time Frame: Baseline, up to Day 9
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MGV354 0.1% | Placebo
Number analyzed (Participants) | 24 | 25
mmHg
  Change from Baseline at 36 hours post Day 7 dose | -1.58 (3.574) | -1.09 (2.209)
  Change from Baseline at 48 hours post Day 7 dose | -1.39 (3.282) | -0.12 (2.541)

4. Secondary Outcome: Part 1: Maximum Observed Concentration [Cmax (ng/mL)]
Description: Based on plasma samples collected at pre-determined nominal time points, dependent on observed concentrations. Approximately 2 mL of venous blood was collected at each time point. Cmax is reported as mass/volume.
Time Frame: Pre-dose, .5, 2, 4, 6, 12, 24, 48, 72, 96, 120 hours post-dose, and Day 7 post-dose
Population: This analysis population includes all subjects who received IP, had at least 1 plasma sample following exposure to non-placebo IP and had no known specimen collection or analytical deviations which would affect the integrity of the data (Pharmacokinetic (PK) Analysis Set). Number Analyzed is the number of subjects with data at visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- MGV354 0.03%: Part 1: MGV354 0.03% ophthalmic suspension, 1 drop in the study eye
- MGV354 0.1%: Part 1: MGV354 0.1% ophthalmic suspension, 1 drop in the study eye
- MGV354 0.3%: Part 1: MGV354 0.3% ophthalmic suspension, 1 drop in the study eye
Arm/Group | MGV354 0.03% | MGV354 0.1% | MGV354 0.3%
Number analyzed (Participants) | 3 | 6 | 6
ng/mL | 0.073 (0.013) | 0.098 (0.032) | 0.327 (0.178)

5. Secondary Outcome: Part 1: Time to Reach Maximum Concentration [Tmax (h)]
Description: Based on plasma samples collected at pre-determined nominal time points, dependent on observed concentrations. Approximately 2 mL of venous blood was collected at each time point.
Time Frame: Pre-dose, .5, 2, 4, 6, 12, 24, 48, 72, 96, 120 hours post-dose, and Day 7 post-dose
Population: PK Analysis Set. Number Analyzed is the number of subjects with data at visit.
Measure: Median (Full Range); unit: hours
Arm/Group | MGV354 0.03% | MGV354 0.1% | MGV354 0.3%
Number analyzed (Participants) | 3 | 6 | 6
hours | 0.483 [0.483 to 23.833] | 0.559 [0.500 to 2.033] | 0.575 [0.567 to 1.983]

6. Secondary Outcome: Part 1: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration [AUClast (ng*h/mL)]
Description: Based on plasma samples collected at pre-determined nominal time points, dependent on observed concentrations. Approximately 2 mL of venous blood was collected at each time point. AUClast is reported as mass*time/volume.
Time Frame: Pre-dose, .5, 2, 4, 6, 12, 24, 48, 72, 96, 120 hours post-dose, and Day 7 post-dose
Population: PK Analysis Set. Number Analyzed is the number of subjects with data at visit.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | MGV354 0.03% | MGV354 0.1% | MGV354 0.3%
Number analyzed (Participants) | 3 | 6 | 6
ng*h/mL | 0.213 (0.336) | 0.157 (0.043) | 1.611 (1.484)

7. Secondary Outcome: Part 1: Area Under the Plasma Concentration-time Curve From Time Zero to 120 Hours Post Dose [AUC0-120 (ng*h/mL)]
Description: Based on plasma samples collected at pre-determined nominal time points, dependent on observed concentrations. Approximately 2 mL of venous blood was to be collected at each time point.
Time Frame: Pre-dose to 120 hours post-dose
Population: Due to the low exposure and the limit of the lower limit of quantitation (LLOQ) (0.05 ng/mL), none of the observed individual profiles could generate valid AUC0-120.
Arm/Group | MGV354 0.03% | MGV354 0.1% | MGV354 0.3%
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From 0 to Infinity [AUCinf (ng*h/mL)]
Description: as for outcome 7
Time Frame: Pre-dose to 120 hours post-dose
Population: Due to the low exposure and the limit of LLOQ (0.05 ng/mL), none of the observed individual profiles could generate valid AUCinf.
Arm/Group | MGV354 0.03% | MGV354 0.1% | MGV354 0.3%
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Part 1: Terminal Elimination Half-life [t1/2 (h)]
Description: as for outcome 7
Time Frame: Pre-dose to 120 hours post-dose
Population: Due to the low exposure and the limit of LLOQ (0.05 ng/mL), none of the observed individual profiles could generate valid t1/2.
Arm/Group | MGV354 0.03% | MGV354 0.1% | MGV354 0.3%
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Part 2: Maximum Observed Concentration [Cmax (ng/mL)]
Description: as for outcome 4
Time Frame: Up to Day 7
Population: PK Analysis Set. Number Analyzed is the number of subjects with data at visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- MGV354 0.03%: Part 2: MGV354 0.03% ophthalmic suspension, next lowest dose from the maximum tolerated dose (MTD) concentration from Part 1, 1 drop in each eye for 7 days
- MGV354 0.1%: Part 2: MGV354 0.1% ophthalmic suspension, MTD concentration determined from Part 1, 1 drop in each eye for 7 days
Arm/Group | MGV354 0.03% | MGV354 0.1%
Number analyzed (Participants) | 6 | 6
ng/mL
  Day 1 | 0.077 (0.026) | 0.139 (0.034)
  Day 7: number analyzed (Participants) | 3 | 5
  Day 7 | 0.132 (0.054) | 0.188 (0.070)

11. Secondary Outcome: Part 2: Time to Reach Maximum Concentration [Tmax (h)]
Description: as for outcome 5
Time Frame: Up to Day 7
Population: PK Analysis Set. Number Analyzed is the number of subjects with data at visit.
Measure: Median (Full Range); unit: hours
Arm/Group | MGV354 0.03% | MGV354 0.1%
Number analyzed (Participants) | 6 | 6
hours
  Day 1 | 0.533 [0.500 to 0.583] | 0.567 [0.550 to 0.583]
  Day 7: number analyzed (Participants) | 3 | 5
  Day 7 | 0.550 [0.483 to 0.550] | 0.533 [0.483 to 1.967]

12. Secondary Outcome: Part 2: Area Under the Concentration-time Curve From 0 to the End of the Dosing Interval Tau [AUCtau (ng*h/mL)]
Description: Based on plasma samples collected at pre-determined nominal time points, dependent on observed concentrations. Approximately 2 mL of venous blood was collected at each time point. AUCtau is reported as mass*time/volume.
Time Frame: Up to Day 7
Population: PK Analysis Set. Number Analyzed is the number of subjects with data at visit.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | MGV354 0.03% | MGV354 0.1%
Number analyzed (Participants) | 2 | 5
ng*h/mL
  Day 1: number analyzed (Participants) | 0 | 1
  Day 1 |  | 0.723 (NA) — Not calculated when only 1 subject analyzed
  Day 7 | 0.392 (0.444) | 1.461 (1.043)

13. Secondary Outcome: Part 2: Accumulation Ratio (Racc)
Description: Accumulation Ratio was derived using Cmax on Day 7 versus Cmax on Day 1. Approximately 2 mL of venous blood was collected at each time point.
Time Frame: Day 7
Population: PK Analysis Set. Number Analyzed is the number of subjects with data at visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MGV354 0.03% | MGV354 0.1%
Number analyzed (Participants) | 3 | 5
ng/mL | 1.893 (1.038) | 1.391 (0.366)

14. Secondary Outcome: Part 3: Observed Concentration at 12 Hours Following Drug Administration [C12 (ng/mL)]
Description: Based on plasma samples collected at pre-determined nominal time points, dependent on observed concentrations. Approximately 2 mL of venous blood was collected at each time point. C12 is reported as mass/volume.
Time Frame: Up to Day 8
Population: PK Analysis Set. Number Analyzed is the number of subjects with data at visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- MGV354 0.1%: Part 3: MGV354 0.1% ophthalmic suspension, MTD concentration determined from Part 2, 1 drop in each eye for 7 days
Arm/Group | MGV354 0.1%
Number analyzed (Participants) | 10
ng/mL
  Day 2: number analyzed (Participants) | 5
  Day 2 | 0.0881 (0.03964)
  Day 8 | 0.1488 (0.11026)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (Part 1: up to 37 days, Part 2: up to 50 days, and Part 3: up to 59 days).
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. This analysis population includes all subjects exposed to investigational product (Safety Analysis Set).
Groups:
- MGV354 0.01% Part 1; MGV354 0.03% Part 1; MGV354 0.1% Part 1; MGV354 0.3% Part 1; Placebo Part 1: 1 drop in the study eye
- MGV354 0.03% Part 2; MGV354 0.1% Part 2; Placebo Part 2; MGV354 0.1% Part 3; Placebo Part 3: 1 drop in each eye for 7 days
Arm/Group | MGV354 0.01% Part 1 | MGV354 0.03% Part 1 | MGV354 0.1% Part 1 | MGV354 0.3% Part 1 | Placebo Part 1 | MGV354 0.03% Part 2 | MGV354 0.1% Part 2 | Placebo Part 2 | MGV354 0.1% Part 3 | Placebo Part 3
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/4 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/4 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 3/6 | 6/6 | 0/8 | 6/6 | 6/6 | 1/4 | 23/25 | 5/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MGV354 0.01% Part 1 (N=6) | MGV354 0.03% Part 1 (N=6) | MGV354 0.1% Part 1 (N=6) | MGV354 0.3% Part 1 (N=6) | Placebo Part 1 (N=8) | MGV354 0.03% Part 2 (N=6) | MGV354 0.1% Part 2 (N=6) | Placebo Part 2 (N=4) | MGV354 0.1% Part 3 (N=25) | Placebo Part 3 (N=25)
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 3 | 6 | 0 | 2 | 6 | 0 | 12 | 1
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 4 | 0 | 2 | 1 | 0 | 7 | 2
Conjunctival cyst (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 7 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 11 | 3
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.